CLINICAL TRIAL: NCT01067937
Title: Multicenter Prospective Study for a Rational Management of Appendicitis in Children
Brief Title: Study for a Rational Management of Appendicitis in Children
Acronym: ALGAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: General Director, Nantes University Hospital, Nantes University Hospital
Masking: None
Other Study IDs: BRD 08/6-L
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Appendicitis
Keywords: Appendicitis; children
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy

INTERVENTIONS:
Procedure: appendectomy — Randomisation will apply to the 8 participating centers as follow: During a first survey period of 6 month, the algorithm is not applied; The six following months, 4 randomised centers applied the algorithm, the others being still survey; The six last month, all centers will apply the algorithm

SUMMARY:
Despite the fact that appendicitis is one of the most frequent surgical pathology in children, its clinical management is still debated. Previous reports have shown rate of appendectomy in children without appendicitis up to 30 %. Morbidity, due to infectious complications or intestinal obstruction, is often between 5 and 10 % of published cases, and increase medical and social costs. Evidence-based medicine concept could therefore be worthwhile in that context, in order to promote rational diagnosis and treatment of that frequent medical condition.An algorithm describing management of children with suspicion of appendicitis was established, based on recent published data, in order to reduce delay between first clinical signs and confirmation of the diagnosis, and to define therapeutic indication such as conservative management and interval appendectomy or patient requiring laparoscopic approach. The main objective of the study is to decrease morbidity and unnecessary appendectomy rates, and secondly to decrease costs, by the use of that algorithm.

ELIGIBILITY:
Inclusion Criteria:

* male and female children, between 4 and 15 years-old, with more than 37,5°C of body temperature during the 3 days before hospital admission, and with abdominal pain located in right or median lower quadrant

Exclusion Criteria:

* children coming from another hospital, children with septic choc, children with co-morbidity in interaction with algorithm (antibiotics allergy, mellitus diabetes, haemostasis disturbance, …)

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 891 (Actual)
Dates: Start 2009-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - WEIL Dominique, Angers
  - DE VRIES Philine, Brest
  - PETIT Thierry, Caen
  - PODEVIN Guillaume, Nantes
  - MCHEIK Jiad, Poitiers
  - AZZIS Olivier, Rennes
  - GARIGNON Cynthia, Saint-Brieuc
  - LARDY Hubert, Tours